CLINICAL TRIAL: NCT00837200
Title: Phase II Pilot Efficacy Trial of the Combination Regimen Oncaspar/Doxil/Decadron (ODD) in Patients With Refractory Lymphoid Malignancies
Brief Title: Oncaspar/Doxil/Decadron in Patients With Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI said to close accrual do to funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Drabick, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-007
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Non-hodgkins Lymphoma; Hodgkins Lymphoma; Multiple Myeloma
Keywords: lymphoma; myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Lymphoma; Neoplasms, Plasma Cell | interventions — pegaspargase; liposomal doxorubicin; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oncaspar, Doxil, Decadron Regimen (Experimental): Once enrolled, patients will receive a cycle (28 days) of Oncaspar (2500 IU/m2 IV on days 1, 15; Doxil 20 mg/m2 IV days 1,15; and Decadron 20 mg PO days 1, 8, 15, 22. Continue until disease progression or unacceptable side effects.
  Interventions: Drug: Oncaspar, Doxil, Decadron

INTERVENTIONS:
Drug: Oncaspar, Doxil, Decadron — Once enrolled, patients will receive a cycle (28 days) of Oncaspar (2500 IU/m2 IV on days 1, 15; Doxil 20 mg/m2 IV days 1,15; and Decadron 20 mg PO days 1, 8, 15, 22. Continue until disease progression or unacceptable side effects.
  Other Names: PEG-asparaginase; PEG-liposomal doxorubicin

SUMMARY:
This is an exploratory study to study the efficacy of combination regimen of Oncaspar/Doxil/Decadron (ODD) in patients with refractory lymphoid malignancies. Patients with any form of lymphoid malignancy will be eligible: acute lymphoblastic leukemia, chronic lymphocytic leukemia, non-Hodgkin's lymphoma, Hodgkin's lymphoma, multiple myeloma and plasma cell leukemia. Patients must have failed standard regimens for their cancers and could have had unlimited number of prior regimens. Patients will be staged appropriately for their disease with clinical examination, laboratory tests, and imaging studies. Both Oncaspar and Doxil will be given on day 1 and 15. Patients will be clinically evaluated prior to each cycle and will have disease assessments every 2 cycles. Responding patients will continue therapy until disease progression or excessive toxicity. Responders who are candidates for allogenic stem cell transplantation could go to conditioning chemotherapy and stem cell transplant after 4 cycles of ODD.

DETAILED DESCRIPTION:
This phase II trial will study the effectiveness of a combination regimen which includes Oncaspar (PEG-asparaginase), Doxil (PEG-liposomal doxorubicin), and Decadron (ODD) in terms of disease response against refractory lymphoid malignancies. Asparaginase is an enzyme that depletes asparagines, a key amino acid for survival and growth of malignant lymphocytes. Its depletion results in death of the neoplastic cell. Asparagine depletion has induced a significant improvement of clinical outcomes in acute lymphoblastic leukemia (ALL) and L-asparaginase has been a mainstay for more than 30 years in the treatment of ALL. Although this drug has been used primarily in ALL, promising results have been reported even in other non-ALL lymphoid malignancies, such as chronic lymphocytic leukemia (CLL), prolymphocytic leukemia, refractory non-Hodgkin's lymphoma (NHL) and multiple myeloma (MM). One of the main goals of this trial is to measure the asparaginase level as a surrogate marker of asparagine depletion with Oncaspar, a PEG-enhanced version of E. coli L-asparaginase. The therapeutic value of the simple, non-pegylated form of L-asparaginase is limited by its short half-life and propensity to cause allergic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented lymphoid malignancies, regardless of their origin (B,T or NK). These include ALL, CLL, HL, NHL, MM and PCL.
* Patients must have failed at least one standard regimen of chemotherapy for their illness. They may have had unlimited prior regimens.
* Performance status of ≤ 2 as per ECOG scale.
* ALT < 2.5 times the upper limit of normal
* Anticipated life expectancy of at least 12 weeks
* Patients will be allowed to have baseline cytopenias, but ANC should be >200/μl and a platelet count > 25,000/ μl (within 2 weeks of starting therapy).
* Patients must have a serum creatinine level ≤ 2 mg/dL (within 2 weeks of starting therapy).
* Male or female adults of at least 18 years of age.
* Signed written informed consent and willingness to meet follow-up schedule and study procedure obligations
* Left Ventricular Ejection Fraction (LVEF) > 40% by echocardiogram or MUGA scan performed within 60 days prior to registration
* Women and men of childbearing potential must agree to employ adequate contraception to prevent pregnancy while on therapy.

Exclusion Criteria:

* Chemotherapy or radiotherapy received within the previous 2 weeks.
* Uncontrolled, active infection requiring IV antibiotics.
* Psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Pregnant or potential for pregnancy.
* Breast-feeding.
* Prior asparaginase therapy complicated by pancreatitis, allergic reaction, hemorrhagic event, or thrombosis
* Previous treatment with pegylated asparaginase
* Prior doxorubicin exposure, more than 400 mg/m2
* Clinically significant CHF
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for at least three years. Prior malignancy is acceptable provided there has been no evidence of disease within the three year interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Drabick, MD, Principal Investigator — Penn State University
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ODD Regimen: Once enrolled, patients will receive a cycle (28 days) of Oncaspar (2500 IU/m2 IV on days 1, 15; Doxil 20 mg/m2 IV days 1,15; and Decadron 20 mg PO days 1, 8, 15, 22. Continue until disease progression or unacceptable side effects.
  Oncaspar, Doxil, Decadron: Once enrolled, patients will receive a cycle (28 days) of Oncaspar (2500 IU/m2 IV on days 1, 15; Doxil 20 mg/m2 IV days 1,15; and Decadron 20 mg PO days 1, 8, 15, 22. Continue until disease progression or unacceptable side effects.
Period: Overall Study
Arm/Group | ODD Regimen
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Oncaspar 2500 IU/m2 D1,15; Doxil 20mg/m2 D1,15; Decadron 20 mg D1,8,15,22
Arm/Group | Treatment
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 64.9 [46 to 80]
Age, Customized [Number; unit: participants]
  Participants over 70 years old | 6
  Partipants under 70 years old | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 13
Participants Diagnosis [Number; unit: participants]
  Multiple Myeloma | 7
  Diffuse Large B-cell Lymphoma | 6
Prior Regimens [Number; unit: participants]
  Pre-Treated with 3 Median prior Regimens | 3
  Not treated with Prior Regimens | 10

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: * Leukemias mainly w/peripheral blood counts/diff every 2 wks/CLL, CT scan before initiation of study, 2nd CT after EOT, no CT at FU
  * Lymphomas restaged w/CT scans of chest/abdomen/pelvis or PET/CT scans after 2 cycles
  * MM monitored w/tumor markers monthly Quantitative immunoglobulins/SPEP w/quantitative M component in MM pts producing full antibody, UPEP w/ quantitative Bence-Jones in MM pts producing only light chains/Serum free light chains obtained all pts/Skeletal surveys at baseline Tumor responses:CR complete resolution of all detectable clinical/radiographic evidence of disease, disappearance of all disease related symptoms, and normalization of biochemical abnormalities for at least 6 wks following treatment and no BM infiltration;PR reduction of all measurable lesions by 50% or more/no new lesions;SD not fulfilling PR criteria/no evidence disease progression;PD increase original tumor mass by more than 25% lesion/new lesion
  * Stable disease > 2mo was a response
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | ODD Regimen
Number analyzed (Participants) | 12
participants | 2

2. Primary Outcome: Study Specific Measure (Response)
Time Frame: 16 Weeks
Measure: Number; unit: participants
Arm/Group | ODD Regimen
Number analyzed (Participants) | 12
participants
  Not Evaluable for Response | 1
  Stable Disease > 2 months | 2
  Progressive Disease | 10

3. Primary Outcome: Study Specific Measure (Number of Participants Taken Off Study)
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | ODD Regimen
Number analyzed (Participants) | 13
participants
  Due to Oncaspar-Related Toxicities | 1
  Not De to Oncaspar-Related Toxicities | 12

ADVERSE EVENTS:
Arm/Group | ODD Regimen
Serious Adverse Events (participants affected / at risk) | 9/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ODD Regimen (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1
Elevated Alk Phos (Metabolism and nutrition disorders) | 1
Elevated AST (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Emboli (Vascular disorders) | 1
Sepsis (Infections and infestations) | 1
Emesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 2 (2)
Infection - unk ANC (Infections and infestations) | 1
Fever (Infections and infestations) | 1
Anorexia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ODD Regimen (N=13)
Decreased WBC (Blood and lymphatic system disorders) | 7
Decreased ANC (Blood and lymphatic system disorders) | 4
Elevated AST (Metabolism and nutrition disorders) | 3
Elevated ALT (Metabolism and nutrition disorders) | 3
Decreased Platelets (Blood and lymphatic system disorders) | 6
Decreased Hemoglobin (Blood and lymphatic system disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes